CLINICAL TRIAL: NCT01035099
Title: A Randomized Open Label Clinical Trial of Fixed Dose Letrozole vs. Titrated Letrozole for In Vitro Fertilization With Cryopreservation of Oocytes and Embryos in Breast Cancer Patients
Brief Title: RCT of Fixed vs Titrated Letrozole in Breast Cancer Patient Undergoing IVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0811010075
Record Dates: First submitted 2009-12-07; First posted 2009-12-18 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Infertility
Keywords: Letrozole; IVF (in vitro fertilization); Cryopreservation; Fertility Preservation; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Titrated dose Letrozole (Experimental): Patients who are randomized to the titrated dose of Letrozole, will start gonadotropins in the evening of day #2 of their menstrual cycle with injectable follicle stimulating hormone (FSH) and human menopausal gonadotropin (HMG). Oral Letrozole will be added to the stimulation in the following titrated regimen.
  Interventions: Drug: Letrozole
- Fixed dose Letrozole (Active Comparator): Patients who are randomized to fixed dose Letrozole will start Letrozole 5mg daily (orally) on the second day of their menstrual cycle and then gonadotropins on the fourth day of their menstrual cycle.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole titrated regimen may be started on day 2 of menstrual cycle:
  Serum Estradiol level <150 pg/ml- No Letrozole; Serum Estradiol Level 150-250 pg/ml- 2.5mg; Serum Estradiol Level 251-350 pg/ml- 5 mg; Serum Estradiol Level >350 pg/ml - 7.5 mg;
  Other Names: Femara- trade name
  Arms: Titrated dose Letrozole
Drug: Letrozole — Fixed dose of 5 mg per day Letrozole will be started on the second day of their menstrual cycle
  Other Names: Femara- trade name
  Arms: Fixed dose Letrozole

SUMMARY:
The purpose of this study is to compare two different ways to administer Letrozole to determine their effectiveness in blocking estrogen production during ovarian stimulation in patients with breast cancer prior to chemotherapy/radiotherapy so that oocytes or embryos can be cryopreserved and patients can possibly achieve a pregnancy after the treatment of breast cancer.

During standard ovulation stimulation, the estrogen levels will exceed normal levels and may reach 10 times the normal level for a 2 week period. This may not be desirable in breast cancer patients. The study hopes to determine if the investigators can stimulate oocyte development in the conventional way and administer different doses of Letrozole as the oocytes develop, to keep estradiol levels low, increase the number of oocytes the investigators are able to recover, and improve the quality of those oocytes.

DETAILED DESCRIPTION:
IVF is a process which involves a schedule of injectable medication to recruit several follicles, each containing an egg, to be retrieved under ultrasound guidance where they can be fertilized. Embryos are then selected to be transferred back into the patient's uterus or are cryopreserved and transferred at a later date.

Letrozole is a potent and highly selective third generation aromatase inhibitor that was developed in the early 1990's. Aromatase is an enzyme of the cytochrome P-450 superfamily and the product of the CYP19 gene, which catalyzes the reaction that converts androgenic substances to estrogens in many tissues, including the granulosa cells of ovarian follicles. Letrozole competitively inhibits the activity of the aromatase enzyme and has a half-life of approximately 48 hours. Because of its potent, sustained suppression in the plasma levels of estradiol, this drug has been recently found to be superior to tamoxifen in the treatment of advanced-stage post-menopausal breast cancer. Conventional ovarian stimulation often results in very high estrogen levels. Since the high estrogen levels are often unsafe for breast cancer patients, fixed dose aromatase inhibitor protocols with Letrozole were developed, to achieve effective ovarian stimulation with reduced estrogen levels to prevent tumor progression and short-term cancer recurrence.

A fixed dose of Letrozole has been used off-label as an ovulation induction agent in many centers to stimulate egg development for infertile couples and patients prior to undergoing chemotherapy for estrogen sensitive cancers.

The purpose of our study is to determine if titrated dose Letrozole in comparison to fixed dose Letrozole during gonadotropin stimulation in IVF in breast cancer patients results in lower estradiol levels and higher mature oocyte yield.

In patients who are scheduled to undergo treatment with IVF for fertility preservation due to breast cancer, we would like to prospectively randomize them to fixed dose vs. titrated dose of Letrozole. Due to time restraints for chemotherapy patients may present for ovarian stimulation prior to Day 2 of their menstrual cycle. If this were to occur, Ganirelix may be started to suppress the pituitary hormones for down regulation prior to starting stimulation medications until day 2 of menstrual bleeding. Eligible subjects will be fully informed about the nature of the trial. Subjects could be enrolled for IVF treatment at any point after breast cancer diagnosis following surgery but before the initiation of chemotherapy, if chemotherapy has been prescribed by their oncologist. After obtaining written informed consent, the subjects will be screened based on inclusion/exclusion criteria, medical and infertility history, Day 2/3 FSH and estradiol, physical and gynecological examination, oncology clearance and the Center's standard screening evaluations for IVF patients. A thorough gynecologic and endocrinologic evaluation will be performed before the start of any treatment. Laboratory assessments will include CBC, chemistry and lipid profile (see attached history and physical form). Vital signs including blood pressure, pulse, and weight will be assessed at baseline (prior to start of stimulation medication), with preoperative evaluation, on day of egg retrieval, and with post retrieval visits.

Patients will have serum blood tests for bHCG, FSH, AMH, Estradiol, and LH and vaginal sonogram on the second day of menstrual bleeding. Start of stimulation medication will proceed only with documentation of a serum negative pregnancy test. Patients will only be eligible to participate in the study for one cycle of in vitro fertilization.

Patients who elect to participate in the study will be provided with gonadotropin medications.

The starting dose of gonadotropins for both study groups would be determined by the patients' age and by antral follicle counts assessed by transvaginal ultrasound at the time of initial consultation. See below:

Age <35 , Antral follicle Count >15 gonadotropin dose 225 IU (150 IU FSH + 75 IU HMG; Age <35, Antral follicle Count <15 gonadotropin dose 300 IU (150 IU FSH + 150 IU HMG; Age 35-39, Antral follicle Count >10 gonadotropin dose 300 IU (150 IU FSH + 150 IU HMG; Age 35-39, Antral follicle Count <10 gonadotropin dose 450 IU (225 IU FSH + 225 IU HMG; Age>40 Independent of antral follicle count, gonadotropin dose 450 IU (225 FSH + 225 IU HMG);

All patients would also be given a daily medication to prevent them from ovulating (Ganirelix), no later than cycle day #7 and continuing until HCG administration.

Group#1-Fixed Letrozole Group: Provided their blood tests and sonograms were within normal limits, patients who are randomized to fixed dose Letrozole will start Letrozole 5mg daily (orally) on the second day of their menstrual cycle and then gonadotropins on the fourth day of their menstrual cycle (Current Letrozole protocol at CRMI). Patients will be monitored with daily blood tests for estradiol and LH and sonogram every 1-3 days. Adjustments to gonadotropin dosing will be made as per usual protocol for IVF. Letrozole dose will not change and will continue for two weeks after egg retrieval.

Group #2-Titrated Letrozole Group: Provided their blood tests and sonograms were within normal limits, patients who are randomized to the titrated dose of Letrozole, will start gonadotropins in the evening of day #2 of their menstrual cycle with injectable follicle stimulating hormone (FSH) and human menopausal gonadotropin (HMG). Oral Letrozole will be added to the stimulation in the following titrated regimen:

Serum Estradiol level <150 pg/ml- No Letrozole; Serum Estradiol Level 150-250 pg/ml- 2.5mg; Serum Estradiol Level 251-350 pg/ml- 5 mg; Serum Estradiol Level >350 pg/ml - 7.5 mg;

The maximal starting dose of Letrozole will be 5 mg, regardless of the initial estradiol level. The Letrozole dose may be reduced if the appropriate suppression of estradiol occurs. The maximal increase or decrease in Letrozole dose will be 2.5 mg/ day. Patients will be monitored with blood tests for estradiol and LH and sonograms starting on the second day of gonadotropin stimulation and every 1-3 days to monitor response and adjust medication dose as per our usual IVF protocol. Letrozole will be stopped for both groups on the day that HCG is given and resumed after egg retrieval. All patients will stay on the same dose of Letrozole that was required for their last day of ovarian stimulation for 2 weeks after stimulation to keep estradiol levels at a minimum. In addition, patients will have serum estradiol levels drawn weekly for 2 weeks after stimulation. Follow-up vital signs will be recorded along with CBC, liver function panel, and cholesterol panel 2 weeks after stimulation. They will also be asked to return 6 months to 1 year after completion of chemotherapy for AMH and FSH levels to evaluate ovarian reserve, and then followed on a yearly basis by phone/mail questionnaire or in person with an annual gynecological examination.

All study patients will be provided with an emergency 24-hour phone number to reach a physician to report adverse reactions to medications, and these physicians will file adverse event report forms to the principal investigator and data safety monitoring board. In addition, they will be asked to report any adverse reactions to medications during follicular monitoring sonograms. All decisions regarding daily medication doses will be determined by the study principal investigator. Otherwise, the treatment of ovarian stimulation, egg retrieval, and cryopreservation is identical to non-study patients undergoing ovarian stimulation, oocyte retrieval, and embryo/oocyte cryopreservation.

Two weeks after retrieval, follow-up instructions will be reviewed. Patients will be advised to refrain from embryo transfer for a minimum of 2 years after chemotherapy. Patients will not be permitted to undergo embryo transfer for a minimum of one year after completing chemotherapy and only after clearance for pregnancy has been obtained from their medical oncologist. Patients will be followed for five years on an annual basis with a follow-up telephone call from one of the investigators inquiring about health status (see patient follow-up data sheet). A pregnancy registry will be created for any pregnancy occurring following enrollment in the study. Detailed pregnancy outcome will be collected between age 2-5 years (see baby follow-up data sheet attached).

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patient with breast cancer diagnosis after surgery and before undergoing chemotherapy desiring fertility preservation with oocyte or embryo cryopreservation
* Healthy subject according to documented medical history and physical examination who has been diagnosed with breast cancer (estrogen and progesterone receptor positive and/or negative)
* Age less that 45 years at time of informed consent
* Verbal or written clearance from medical or surgical oncologist to undergo controlled ovarian hyperstimulation-IVF
* Delay to chemotherapy treatment will not jeopardize cancer treatment outcome
* Ovarian stimulation will not affect cancer treatment plan
* Transvaginal ultrasound scan (US) within one month of starting stimulation with no clinically significant pelvic mass
* Serum FSH level (Day 2-4) less than 25
* Negative pregnancy test prior to beginning Letrozole or gonadotropin therapy
* Willing and able to comply with the protocol
* Voluntary provision of written informed consent, prior to any study related procedure that was not part of normal medical care, with the understanding that the subject can withdraw consent at any time without prejudice to her future medical care
* Willingness to provide follow-up information on herself and babies born as part of this study

Exclusion Criteria:

* Patients not medically cleared by their oncologist
* Patients with stage IV breast cancer based on the poor prognosis, general health of the patient, and higher uncertainty with delaying chemotherapy
* Any clinically relevant abnormal laboratory value (FSH >25 miu/ml, renal function, (greater than two times normal value), hepatic function (greater than two times normal value), blood biochemistry, hematology (elevated white blood count greater than 1.5 times the normal value, hemoglobin <10mg/dL, thrombocytopenia), abnormal cholesterol profile (total cholesterol ≥ 300mg/dL, abnormal LDL greater than 2 times normal value,) based on a fasting sample during the screening phase
* Contraindications for the use of gonadotropins (i.e. Tumors other than breast cancer, pregnancy, lactation, undiagnosed vaginal bleeding)
* Recent or current medical conditions where the patient is not medically stable to undergo stimulation or egg retrieval, HIV infection, diabetes, cardiovascular disease, gastrointestinal, hepatic disease, undiagnosed pelvic mass, renal or pulmonary disease
* History or presence of alcohol or drug abuse within 12 months of signing consent
* History of severe allergic or anaphylactic reactions or hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol
* Administration of investigational drugs within three months prior to signing the informed consent
* Use of insulin sensitizing agents at least one month prior to signing informed consent
* Any patient who is not a candidate for IVF

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, MD, Principal Investigator — Weill Cornell Medical Cornell
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine — http://www.ivf.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 subjects were enrolled; One subject 1 later withdrew consent prior to randomization.
Groups:
- Titrated Dose Letrozole: Patients who are randomized to the titrated dose of Letrozole, will start gonadotropins in the evening of day #2 of their menstrual cycle with injectable follicle stimulating hormone (FSH) and human menopausal gonadotropin (HMG). Oral Letrozole will be added to the stimulation in the following titrated regimen.
  Letrozole: Letrozole titrated regimen may be started on day 2 of menstrual cycle:
  Serum Estradiol level <150 pg/ml- No Letrozole; Serum Estradiol Level 150-250 pg/ml- 2.5mg; Serum Estradiol Level 251-350 pg/ml- 5 mg; Serum Estradiol Level >350 pg/ml - 7.5 mg;
Period: Overall Study
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 41 subjects were enrolled; One subject 1 later withdrew consent prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 22 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 21 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mature Oocyte Yield
Description: Mature oocyte yield in each group
Time Frame: 1 to 2 months
Population: Only 39 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization; 1 subject in the Fixed dose group had no oocytes harvested, so this measure could not be calculated for that patient).
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 21
oocytes | 5.1 (8.4) | 7.9 (8.2)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.31, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

2. Primary Outcome: Percent of Mature Oocyte Yield
Description: The percentage of mature oocyte obtained will be compared from both arms. Calculated as number of mature oocytes divided by number of oocytes retrieved (per patient).
Time Frame: 1 to 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of mature oocytes
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 21
percentage of mature oocytes | 0.29 (0.38) | 0.46 (0.41)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.19, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

3. Secondary Outcome: Participant Cycle Cancellation Rate
Description: Cycle cancellation rate- participant
Time Frame: 1 to 2 months
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Breast Cancer Recurrence Rate
Description: 5 year follow-up breast cancer recurrence rate
Time Frame: 5 years
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Peak Serum Estradiol Level
Description: Peak Serum Estradiol Level (pg/ml)
Time Frame: 1 to 2 months
Population: Only 40 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization).
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 22
pg/ml | 603.1 (213.4) | 771.1 (401.1)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.12, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

6. Secondary Outcome: FSH ng/ml (Cycle Day 2)
Description: FSH ng/ml on Cycle Day 2
Time Frame: 1 to 2 months
Population: Only 37 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization; Three subjects in Titrated group did not have FSH recorded).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 15 | 22
ng/ml | 5.9 (2.0) | 5.8 (1.6)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.77, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

7. Secondary Outcome: AMH ng/ml (Cycle Day 2)
Description: AMH ng/ml on Cycle Day 2
Time Frame: 1 to 2 months
Population: Only 33 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization; Three subjects in Titrated group did not have AMH recorded and 4 patients in the Fixed group did not have AMH recorded).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 15 | 18
ng/ml | 2.1 (1.6) | 2.4 (1.4)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.63, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

8. Secondary Outcome: AF Count
Description: Antral follicle count
Time Frame: 1 to 2 months
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Total Days Stimulation Medications
Description: Total days of stimulation medications
Time Frame: 1 to 2 months
Population: Only 40 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 22
days | 10.1 (1.7) | 11.2 (2.7)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.14, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

10. Secondary Outcome: Total Medication Dose
Description: Total medication dose given
Time Frame: 1 to 2 months
Population: Only 40 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization).
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 22
mg | 34.0 (7.0) | 55.3 (14.3)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p < 0.0001, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

11. Secondary Outcome: Total Number of Oocytes
Description: Total number of oocytes retrieved
Time Frame: 1 to 2 months
Population: Only 40 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization).
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 22
oocytes | 17.1 (10.3) | 19.0 (11.2)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.58, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

12. Secondary Outcome: Number of Follicles on Day of HCG
Description: Number of follicles on day of Human Chorionic Gonadotrophin (HCG)
Time Frame: 1 to 2 months
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Fertilized Oocytes
Description: Number of fertilized oocytes among participants
Time Frame: 1 to 2 months
Population: Only 39 subjects analyzed of 41 (1 subject later withdrew consent prior to randomization; One subject in Fixed group did not have this information recorded).
Measure: Mean (Standard Deviation); unit: fertlized oocytes
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 18 | 21
fertlized oocytes | 3.7 (5.8) | 5.3 (6.4)
Statistical Analysis 1: Comparison: Titrated Dose Letrozole vs Fixed Dose Letrozole; Test type: Superiority; p = 0.42, t-test, 2 sided; Nonparametric Wilcoxon rank-sum test confirmed these results

14. Secondary Outcome: Number of Good Quality Embryos
Description: Number of good quality embryos among participants
Time Frame: 1 to 2 months
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Breast Cancer Recurrence at Year 1-2
Description: Number of Subjects with Breast Cancer Recurrence at Year 1-2
Time Frame: 1 to 2 years
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Breast Cancer Recurrence at Year 2-3
Description: Number of Subjects with Breast Cancer Recurrence at year 2-3
Time Frame: 2- 3 years
Population: This information was not recorded.
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Only 40 subjects analyzed out of 41 (1 subject was not included because they withdrew consent prior to randomization).
Arm/Group | Titrated Dose Letrozole | Fixed Dose Letrozole
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 6/18 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titrated Dose Letrozole (N=18) | Fixed Dose Letrozole (N=22)
abdominal pain (Gastrointestinal disorders) | 6 (6) | 4 (4)
OHSS (Reproductive system and breast disorders) | 2 (2) | 1 (1) — Ovarian hyperstimulation syndrome

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT01035099/Prot_SAP_000.pdf